CLINICAL TRIAL: NCT00733083
Title: A Comparative Study With Pre-Emptive Parenteral Oxycodone, Morphine and Dexamethasone in the Treatment of Postoperative Pain in Paediatric Patients 4 to 12 Years of Age
Brief Title: A Comparative Study With Parenteral Oxycodone, Morphine and Dexamethasone in Postoperative Pain in Paediatric Patients
Acronym: DOM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Turku (Other)
Responsible Party: MD, PhD Tuula Manner, Turku university hospital, Finland
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DOM
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Last update posted 2008-08-12 (Estimated); Status verified 2008-08

CONDITIONS: Post Tonsillectomy Pain
Keywords: tonsillectomy; paediatric; pain; child; opiates; pre-emptive; oxycodone; morphine; dexamethasone
MeSH Terms: conditions — Pain | interventions — Morphine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): 0,1 mg/kg of oxycodone
  Interventions: Drug: 0,1 mg/kg of oxycodone
- 2 (Active Comparator): 0,1 mg/kg of morphine
  Interventions: Drug: Morphine 0,1 mg/kg
- 3 (Active Comparator): 0,5 mg/kg dexamethasone (max 24 mg
  Interventions: Drug: Dexamethasone 0,5 mg/kg
- 4 (Placebo Comparator): NaCl 0,9%
  Interventions: Drug: NaCl 0,9%

INTERVENTIONS:
Drug: 0,1 mg/kg of oxycodone — solution for injection, 0,1 mg/kg, one injection in the beginning of anesthesia
  Other Names: Oxynorm
  Arms: 1
Drug: Morphine 0,1 mg/kg — solution for injection, 0,1 mg/kg, one injection in the beginning of anesthesia
  Other Names: Morphin
  Arms: 2
Drug: Dexamethasone 0,5 mg/kg — solution for injection, 0,5 mg/kg, one injection in the beginning of anesthesia
  Other Names: Oradexon
  Arms: 3
Drug: NaCl 0,9% — solution for injection one injection in the beginning of anesthesia
  Other Names: NaCl 0,9% Braun
  Arms: 4

SUMMARY:
The aim of this randomized, double-blind study is to compare parenteral pre-emptive oxycodone, morphine and dexamethasone with placebo in the treatment of postoperative pain in paediatric patients 4 to 12 years of age. The investigators hope to find out whether there are any differences in postoperative pain and/or adverse effects among these groups.

DETAILED DESCRIPTION:
After the induction of anaesthesia and before intubation the child receives one of the research drugs in a double-blind fashion: 0.1 mg/kg of oxycodone , 0.1 mg/kg of morphine, 0.5 mg/kg dexamethasone (max 24 mg), or placebo. All the research drugs are diluted into a dose of 10 ml with NaCl 0.9%, the placebo being solely the dilute.

The patients are followed minimum 4h postoperatively: first in the recovery room, and after the patient is stable enough the study is continued in the day-patient unit. Level of pain and adverse effects are registered all on same predetermined intervals being 15 min during the first postoperative hour, followed by interval of 30 min until the discharge.

The safety measurements noted include pulse, respiratory rate, non-invasive blood pressure and peripheral oxygen saturation are recorded on the same intervals The registering of pain, adverse effects and given medication continues at home for 48 hours post operatively with a questionnaire filled by the parents.

ELIGIBILITY:
Inclusion Criteria:

* 4 to 12 years of age
* Scheduled to tonsillectomy
* ASA class I or II
* Written informed consent is obtained from the parents and the child (when appropriate).

Exclusion Criteria:

* Allergy to morphine, oxycodone or dexamethasone

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
The difference of needed rescue pain medication post operatively | predetermined intervals being 15 min during the first postoperative hour, followed by interval of 30 min for 4 first postop hours. At home pain and adverse effects are registered by parent at 24 hours and 48 hours.

SECONDARY OUTCOMES:
differences in adverse effects | In hospital 4 hours with first hour in 15 min intervals, then 30 min. At home 24+48h

CONTACTS AND LOCATIONS:
Overall Officials: Tuula Manner, MD, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University hospital, Turku, Finland